CLINICAL TRIAL: NCT04340557
Title: Randomized Open Label Study of Standard of Care Plus an Angiotensin II Receptor Blocker Compared to Standard of Care Alone to Minimize the Progression to Respiratory Failure in SARS-CoV-2 Infection
Brief Title: Do Angiotensin Receptor Blockers Mitigate Progression to Acute Respiratory Distress Syndrome With SARS-CoV-2 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Matthew Geriak, Investigational Pharmacist, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVID-ARB; 2003902 (Other: Sharp HealthCare Institutional Review Board (SHC IRB))
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV Infection
Keywords: Coronavirus; Angiotensin receptor blocker; SARS-CoV-2; COVID-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections; COVID-19 | interventions — Losartan; Standard of Care

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of two groups: Standard of Care or Standard of Care plus an ARB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Study drug+SOC) (Experimental): Standard of Care plus an ARB to be taken orally twice daily for up to 10 days or until discharged from the hospital, whichever occurs first. Investigator may increase dose on days 2 - 10 if confident the subject will tolerate.
  Interventions: Drug: Losartan
- Group B (SOC) (No Intervention): Standard of Care

INTERVENTIONS:
Drug: Losartan — Standard of care plus the starting dose of losartan 12.5mg (investigator has option to increase dose on days 2-10 based on tolerance of SBP) of losartan taken twice daily for up to 10 days. Upon the treating clinician's discretion, losartan may be continued beyond 10 days for non-COVID-19 indications.
  Other Names: Losartan + Standard of Care
  Arms: Group A (Study drug+SOC)

SUMMARY:
The purpose of this research is to identify whether or not Angiotensin Receptor Blockers (ARB) can halt the progression to respiratory failure requiring transfer into the intensive care unit (ICU), as well as halt mechanical ventilation in subjects with mild to moderate hypoxia due to the corona virus that causes COVID-19. Based on previous animal studies, the researchers hypothesize that the addition of an ARB is beneficial in abating acute lung injury in subjects in early stages of SARS-CoV-2 viral induced hypoxia.

DETAILED DESCRIPTION:
This is an investigator initiated, open label, multicenter, two arm, randomized study to compare the impact of adding an ARB to the Standard of Care (SOC) to the SOC without an ARB. Randomization ratio will be 1:1. The goal of this study is to identify whether or not ARBs have an impact on inhibiting the progression to respiratory failure requiring mechanical ventilation in patients with mild to moderate hypoxia in the setting of COVID-19. The addition of an ARB to the standard of care treatment for these patients may be beneficial in abating acute lung injury in patients in early stages of SARS-CoV-2 induced hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 positive test result
* Mild to moderate respiratory symptoms of COVID-19.
* Systolic blood pressure ≥ 105 mmHg.
* Screen within 3 days of a positive COVID-19 test.
* Age ≥18 years old.
* Access to a phone in the hospital room or an electronic device that is capable of receiving phone or video calls.
* Able to read/write/speak English or Spanish fluently.
* Subjects must have the capacity to provide consent or an appropriate LAR to provide informed consent.
* Negative pregnancy test for women of childbearing potential and subject is randomized to the study arm.

Exclusion Criteria:

* Severe allergy to any ARB or ACE-inhibitor, including angioedema
* In the intensive care unit at screening.
* Home meds include any kind of ACE inhibitor or ARB
* Acute Kidney Injury (50% reduction in GFR from baseline at admission to any time during treatment in the study treatment arm)
* Hyperkalemia >5.0 mmol/L at baseline or any time during treatment in the study treatment arm
* Creatinine Clearance < 30 ml/min at baseline or any time during treatment in the study treatment arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Geriak, PharmD, Study Director — Sharp HealthCare
Locations (3):
- United States (3):
  - Sharp Grossmont Hospital, La Mesa, California
  - Sharp Chula Vista Medical Center, San Diego, California
  - Sharp Memorial Hospital, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geriak M, Haddad F, Kullar R, Greenwood KL, Habib M, Habib C, Willms D, Sakoulas G. Randomized Prospective Open Label Study Shows No Impact on Clinical Outcome of Adding Losartan to Hospitalized COVID-19 Patients with Mild Hypoxemia. Infect Dis Ther. 2021 Sep;10(3):1323-1330. doi: 10.1007/s40121-021-00453-3. Epub 2021 May 11. PMID 33977506

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan + Standard of Care: Standard of Care plus an ARB to be taken orally twice daily for up to 10 days or until discharged from the hospital, whichever occurs first. Investigator may increase dose on days 2 - 10 if confident the subject will tolerate.
  Losartan: Standard of care plus the starting dose of losartan 12.5mg (investigator has option to increase dose on days 2-10 based on tolerance of SBP) of losartan taken twice daily for up to 10 days.
- Standard of Care: Patient will receive the hospital Standard of Care for their condition
Period: Overall Study
Arm/Group | Losartan + Standard of Care | Standard of Care
Started | 16 | 15
Completed | 15 | 13
Not Completed | 1 | 2
Not completed — Transferred to ICU and/or death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group A (Study Drug+SOC): Standard of Care plus an ARB to be taken orally twice daily for up to 10 days or until discharged from the hospital, whichever occurs first. Investigator may increase dose on days 2 - 10 if confident the subject will tolerate.
  Losartan: Standard of care plus the starting dose of losartan 12.5mg (investigator has option to increase dose on days 2-10 based on tolerance of SBP) of losartan taken twice daily for up to 10 days.
- Total: Total of all reporting groups
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC) | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [33 to 95] | 54.9 [23 to 91] | 57.1 [23 to 95]
Age, Continuous [Median (Full Range); unit: years] | 54 [33 to 95] | 53 [23 to 91] | 53 [23 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 2 | 3
  Black/African America | 1 | 0 | 1
  Hispanic | 12 | 13 | 25
  Asian | 0 | 0 | 0
  Unknown | 2 | 0 | 2
Days from Hospital Admission to Enrollment [Median (Full Range); unit: days] | 2 [1 to 6] | 2 [1 to 5] | 2 [1 to 6]
Charlson Comorbidity Index [Mean (Full Range); unit: scores on a scale] — The revised Charlson Comorbidity Index is a weighted index to predict risk of death within 10 yrs for patients with specific comorbid conditions. 17 conditions were included in the revised index. Each condition was assigned from 0 to 6 and were summed to produce the score (https://www.mdcalc.com/charlson-comorbidity-index-cci) The lowest to highest possible score is 0 to 102. The higher the score indicates the higher probability of mortality. This scale was utilized to illustrate the clinical similarity between the two groups at baseline.
  scores on a scale | 2.06 [0 to 6] | 1.87 [0 to 5] | 1.97 [0 to 6]
Comorbidities [Count of Participants; unit: Participants]
  Diabetes mellitus | 3 | 5 | 8
  Hypertension | 7 | 5 | 12
  Obesity (BMI >/= 30 kg/m^2) | 8 | 5 | 13
  Tobacco Use | 4 | 2 | 6
  Cardiovascular Disease | 1 | 0 | 1
Receipt of Concomitant SARS-CoV-2 Medications [Count of Participants; unit: Participants]
  Remdesivir | 4 | 5 | 9
  Glucocorticoids > 2 doses | 2 | 5 | 7
  Azithromycin | 2 | 3 | 5
  Hydroxychloroquine | 2 | 1 | 3
  Convalescent Plasma | 1 | 1 | 2
  Anti-thrombotics | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Ventilation
Description: Number of subjects requiring transfer into ICU for mechanical ventilation due to respiratory failure
Time Frame: from date of patient admission to date of patient discharge or date of death, whichever came first, assessed up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 16 | 15
Participants | 1 | 1

2. Secondary Outcome: ICU Transfer
Description: Number of subjects transferred from non-ICU bed to an ICU bed
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 16 | 15
Participants | 1 | 2

3. Secondary Outcome: Oxygen Therapy
Description: Mean number of liters of oxygen consumed
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: liters
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 16 | 15
liters | 10,469 [0 to 49,968] | 82,734 [0 to 748,984]

4. Other Pre Specified Outcome: Length of Hospital Stay
Description: Length of hospital stay from admission to discharge
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: days
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 16 | 15
days | 9 [3 to 30] | 10 [3 to 34]

5. Other Pre Specified Outcome: In Hospital Mortality
Description: Number of subjects who expired while hospitalized
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 16 | 15
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From enrollment into the study until hospital discharge or death, assessed up to 45 days.
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 3/16 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Study Drug+SOC) (N=16) | Group B (SOC) (N=15)
Hypotension (SBP<100) (Vascular disorders) | 3 (3) | 4 (4)
Body aches (General disorders) | 1 (1) | 1 (1)
Cough (General disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 0 (0) | 2 (2)
Transaminitis (General disorders) | 1 (1) | 1 (1)
Malnutrition (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The generalizability is limited by small size of the study population, unblinded design, and all the subjects being screened from three hospitals in close proximity in one geographic area in Southern California.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT04340557/Prot_SAP_000.pdf